CLINICAL TRIAL: NCT00557531
Title: Safety and Feasibility of the Injectable BL-1040 Implant
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioLineRx, Ltd. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: BioLineRx, Public Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1040.01; 1040.01
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BL-1040 (Experimental)
  Interventions: Device: BL-1040

INTERVENTIONS:
Device: BL-1040 — 2 mL of BL-1040

SUMMARY:
This is a Phase I, multi-center, open label study designed to assess the safety and feasibility of the injectable BL-1040 implant to provide scaffolding to infarcted myocardial tissue.

DETAILED DESCRIPTION:
ENDPOINTS Preliminary safety endpoints Occurrence of all adverse events including but not limited to All MIs Cardiovascular hospitalization

Serious ventricular arrhythmias sustained:

VT (symptomatic or sustained VT [duration longer than 30 seconds or 100 beats, or associated with hemodynamic collapse]) VF symptomatic bradycardia, pauses of longer than 3.0 seconds, complete atrioventricular block, Mobitz II atrioventricular block Symptomatic heart failure (NYHA criteria + physical examination OR hospitalization due to heart failure) Renal failure Stroke Death

Secondary safety endpoints Change from baseline in LV dimensions (end-systolic volume index, end-diastolic volume index) Change from baseline in regional (infarct related) and global wall motion score Change from baseline in ejection fraction Cardiac rupture NT-proBNP

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 to 75 years of age, inclusive
* Male or female
* Negative pregnancy test for women of child-bearing potential, or surgically sterile, or post menopausal
* Acute MI defined as:

  * Typical rise and gradual fall (troponin) or more rapid rise and fall (CK-MB) of biochemical markers of myocardial necrosis with at least one of the following:

    * Ischemic symptoms;
    * Development of pathologic Qwaves on the ECG;
    * ECG changes indicative of ischemia (ST segment elevation or depression)
    * First anterior or inferolateral STEMI or Qwave MI (QMI Anterior: V1-V3 or V1-V4 or V1-V5 or V1-V6.QMI Inferior: L2, L3, AVF, or L2, L3, AVF+ V5, V6 or L2, L3, AVF+ V6-V9 [posterior leads])
    * Regional wall motion score index (at least 4 out of 16 akinetic segments)
* One or more of the following:

  * LVEF >20% and <45% measured and calculated by 2-dimensional measurement
  * Biomarkers: peak CK > 2000 IU
  * Infarct size > 25% as measured by MRI
  * Successful revascularization with PCI with 1 stent only, within 7 days of the index MI
  * At time of application of study device, patient must have patent infarct related artery (IRA) and TIMI flow grade = 3

Exclusion Criteria:

* History of CHF, Class I to Class IV, as per NYHA criteria
* History of prior LV dysfunction
* At time of application of study device - Killip III-IV (pulmonary edema, cardiogenic shock - hypotension systolic < 90 mmHg and evidence of peripheral hypoperfusion oliguria, cyanosis, sweating) or HR > 100 bpm
* Prior CABG
* Prior MI
* History of stroke
* Significant valvular disease (moderate or severe)
* Patient is a candidate for CABG or PCI on non-IRA
* Patient is being considered for CRT within the next 30 days
* Renal insufficiency (eGFR < 60)
* Chronic liver disease (> 3 times upper limit of normal)
* Life expectancy < 12 months
* Current participant in another clinical trial, or participation in another trial within the last 6 months
* Any contraindication to coronary angiography, MRI or PCI procedures
* Patient taking anti-coagulation medication prior to MI
* Pregnant or lactating women; pregnancy confirmed by urine pregnancy test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all AEs including but not limited to All MIs CV hospitalization Serious ventricular arrhythmias sustained: Symptomatic heart failure Renal failure Stroke Death | 6 months

SECONDARY OUTCOMES:
Change from baseline in LV dimensions (end-systolic volume index, end-diastolic volume index) Change from baseline in regional (infarct related) and global wall motion score Change from baseline in ejection fraction Cardiac rupture NT-proBNP | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Vermeersch, MD, Principal Investigator — Antwerp MC
Locations (1):
- Heidelberg University MC, Heidelberg, Germany